CLINICAL TRIAL: NCT00999232
Title: Assess the Effect of Erythromycin on the Rate of Success in Placement of a Self-propelled Feeding Tube
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canisius-Wilhelmina Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bengmark_v1
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2009-10

CONDITIONS: Pancreatitis
Keywords: erythromycin; prokinetics; nasojejunal tubes; Bengmark feeding tube; post-pyloric feeding; pancreatitis; Non-critically ill patients having pancreatitis who require jejunal enteral nutrition
MeSH Terms: conditions — Pancreatitis | interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Erythromycin (Experimental)
  Interventions: Drug: Erythromycin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythromycin — Subjects receive 4x250mg erythromycin i.v. daily after intubation of a self-propelled feeding tube
  Arms: Erythromycin
Drug: Placebo — Subjects receive 4x placebo i.v. daily after intubation of a self-propelled feeding tube
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of erythromycin on the Rate of Success in Placement of a Self-propelled Feeding Tube.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Having pancreatitis
* Require jejunal enteral nutrition

Exclusion Criteria:

* Known impaired peristalsis (critically ill patients, postoperative patients, history of surgery of the stomach/duodenum)
* Pregnancy
* Hypersensibility to erythromycin
* Cardiac arrhythmias with a prolonged QT-time
* Simultaneous usage of drugs impairing peristalsis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The success rate of spontaneous positioning the tubes tip into the jejunum, beyond Treitz ligament, after 48 hours.

SECONDARY OUTCOMES:
The success rate of spontaneous positioning the tubes tip into the jejunum, beyond Treitz ligament, after 24 hours.
Adverse events using this self-propelled tube

REFERENCES:
- [Derived] van den Bosch S, Witteman E, Kho Y, Tan AC. Erythromycin to promote bedside placement of a self-propelled nasojejunal feeding tube in non-critically ill patients having pancreatitis: a randomized, double-blind, placebo-controlled study. Nutr Clin Pract. 2011 Apr;26(2):181-5. doi: 10.1177/0884533611399924. PMID 21447772